CLINICAL TRIAL: NCT02729935
Title: Efficacy and Tolerance of Parecoxib for Prevention of Catheter-related Bladder Discomfort in Patients Undergoing Catheterization After TURBT: A Prospective, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Parecoxib for Treatment of Catheter Related Bladder Discomfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ali JENDOUBI, MD, Assistant Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: University Of Tunis El Manar
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Pain
Keywords: Parecoxib; Bladder Discomfort
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parecoxib (Experimental): 40 mg of intravenous parecoxib (DYNASTAT )30 min before surgery
  Interventions: Drug: Parecoxib
- Placebo (Placebo Comparator): An equal volume of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parecoxib — 40 mg of intravenous parecoxib 30 min before surgery
  Other Names: DYNASTAT
  Arms: Parecoxib
Drug: Placebo — An equal volume of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Catheter-related bladder discomfort (CRBD) is defined as an urge to void or discomfort in the supra-pubic region; reported postoperatively in patients who have had urinary catheterization intra-operatively. In the present study, the investigators evaluated Parecoxib (P) for preventing CRBD in patients undergoing catheterization after transurethral resection of bladder tumor (TURBT).

DETAILED DESCRIPTION:
Participants will be randomized into one of two study groups: Group P: 40 mg of intravenous parecoxib 30 min before surgery and Control Group C: an equal volume of saline.

Lumber subarachnoid block was administered with 2 ml 0.5% hyperbaric bupivacaine and 2.5 µg Sufentanyl. Intra-operatively, urinary catherization was performed with a 16 Fr Foley's catheter, and the balloon was inflated with 10 ml distilled water. The CRBD was assessed at 0, 1, 2, and 6 h after patient's arrival in the post-anaesthesia care unit. Severity of CRBD was graded as none, mild, moderate and severe.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/=18)
2. Male or female
3. Undergoing catheterization after transurethral resection of bladder tumor (TURBT)
4. Under spinal anesthesia
5. Subject is American Society of Anesthesiologists (ASA) physical status 1 or 2.

Exclusion Criteria:

1. Patient who disagrees to participate this investigation
2. Patient with severe cardiovascular disease
3. Patient with small-sized foley catheter (less than 18 Fr.)
4. Patinets with bladder outflow obstruction
5. Patient with overactive bladder (frequency >3 times,in the night or >8 times in 24 h)
6. Patients with chronic renal failure
7. Patient with morbid obesity
8. Patient with medications for chronic pain
9. Patient with disturbance of the central nervous system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reducing of Catheter related bladder discomfort symptoms | at postoperatively 30th minutes, 1st, 2nd, 4th, 6th and 12th hours
  CRBD was evaluated with a 4 point scale (1; no discomfort, 2; mild, revealed on questioning only, 3; moderate, stated by the patient without questioning, 4; severe, urinary urgency executed by behavioral responses, such as attempts to remove urinary catheter, restless extremity movements, verbal responses) at postoperatively 30th minutes, 1st, 2nd, 4th, 6th and 12th hours.

SECONDARY OUTCOMES:
Severity of Pain at suprapubic area | at postoperative 0, 1, 6 and 12 hours
  Assessed by Visual Analogue Scale (VAS) and rescue analgesia requirement ( Paracetamol or nefopam)
safety and tolerability of parecoxib | During the first 24 hours
  Blood loss, length of hospitalization, renal function and postoperative cardiovascular (CV) events

CONTACTS AND LOCATIONS:
Overall Officials: Ali JENDOUBI, Principal Investigator — University Tunis El Manar
Locations (1):
- Ali JENDOUBI, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jendoubi A, Aissi W, Abbes A, Bouzouita A, Fourati S, Necib H, Ghedira S, Houissa M. Efficacy and safety of Parecoxib for prevention of catheter-related bladder discomfort in patients undergoing transurethral resection of bladder tumor: Prospective randomised trial. Indian J Anaesth. 2018 Jun;62(6):461-465. doi: 10.4103/ija.IJA_137_18. PMID 29962529